CLINICAL TRIAL: NCT04906590
Title: Assessment of Brain Tau Burden in Participants With Parkinson's Disease in the PPMI Study (PPMI Tau PET Imaging)
Brief Title: PPMI Tau PET Imaging
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Michael J. Fox Foundation for Parkinson's Research (Other)
Collaborators: Institute for Neurodegenerative Disorders (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: PPMI-008
Record Dates: First submitted 2021-05-13; First posted 2021-05-28 (Actual); Last update posted 2023-04-21 (Actual); Status verified 2023-04

CONDITIONS: Parkinson Disease
MeSH Terms: conditions — Parkinson Disease | interventions — ((18)F)PI-2620

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Study Drug (Experimental): All participants will receive PI-2620.
  Interventions: Drug: [18F] PI-2620

INTERVENTIONS:
Drug: [18F] PI-2620 — Evaluation of the radiopharmaceutical imaging agent PI-2620 in detecting TAU brain burden.

SUMMARY:
The Assessment of Brain Tau Burden in Participants with Parkinson's Disease in the PPMI Study (PPMI Tau PET Imaging) will evaluate if [18F] PI-2620 facilitates better understanding of Tau deposition in the brain in Parkinson's disease (PD).

DETAILED DESCRIPTION:
The Assessment of Brain Tau Burden in Participants with Parkinson's Disease in the PPMI Study (PPMI Tau PET Imaging) is a companion study to the Parkinson's Progression Markers Initiative Clinical protocol (PPMI-002; NCT04477785). After consenting to the PPMI Clinical protocol, participants interested in completing an additional scan under this study will be asked to complete consent, additional activities, and one [18F]PI-2620 PET imaging scan as part of this study. Enrollment in the PPMI Tau PET Imaging companion study will facilitate comparison of tau deposition to clinical, imaging, blood and CSF tau already acquired in these PPMI participants under the PPMI Clinical protocol. The primary goal of this imaging study is to test whether positron emission tomography (PET) with [18F] PI-2620 can visualize in vivo brain tau deposition in participants with PD. The secondary goal is to evaluate tau deposition in PD LRRK2 mutation carriers given recent data that tau pathology may be present in those individuals.

ELIGIBILITY:
Inclusion Criteria:

* Enrolled in PPMI Clinical protocol
* Able to provide informed consent
* Male or Female (Females must meet additional criteria specified below, as applicable)

  * Females must be of non-childbearing potential or using a highly effective method of birth control 14 days prior to until at least 24 hours after injection of [18F]PI-2620.
  * Non-childbearing potential is defined as a female that must be either postmenopausal (no menses for at least 12 months prior to PET scan) or surgically sterile (bilateral tubal ligation, bilateral oophorectomy or hysterectomy).
  * Highly effective method of birth control is defined as practicing at least one of the following: A birth control method that results in a less than 1% per year failure rate when used consistently and correctly, such as oral contraceptives for at least 3 months prior to injection, an intrauterine device (IUD) for at least 2 months prior to injection, or barrier methods, e.g., diaphragm or combination condom and spermicide. Periodic abstinence (e.g. calendar, ovulation, symptothermal, post-ovulation methods) is not acceptable.
  * Females of childbearing potential must not be pregnant, breastfeeding or lactating.
  * Females of childbearing potential have a negative urine pregnancy test prior to [18F]PI-2620 injection on day of PET scan.

Exclusion Criteria:

* Exposure to an effective radiation dose of 50 mSv, which would be above the acceptable annual limit established by the US Federal Guidelines during the past year.
* Any other medical or psychiatric condition or lab abnormality, which in the opinion of the Site Investigator might preclude participation.

Ages: 30 Years to 100 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 23 (Actual)
Dates: Start 2021-08-30 (Actual); Primary Completion 2023-01-30 (Actual); Study Completion 2023-02-01 (Actual)

PRIMARY OUTCOMES:
Determination of [18F]PI-2620 standard uptake value ratio (SUVR) targeting brain tau deposition in comparison between Parkinson disease and healthy control participants. | 90 minutes

CONTACTS AND LOCATIONS:
Locations (1):
- Institute for Neurodegenerative Disorders, New Haven, Connecticut, United States